CLINICAL TRIAL: NCT06214377
Title: Effects of Transcranial Direct Current Stimulation (tDCS) on Pain Modulation in Individuals With Parkinson's Disease in the Off State
Brief Title: Transcranial Direct Current Stimulation for Treating Parkinson´s Disease-related Pain in OFF State
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Collaborators: Universidad Rey Juan Carlos (Other); Hospital Beata María Ana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ParkOFF-tDCS
Record Dates: First submitted 2023-11-29; First posted 2024-01-19 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-06

CONDITIONS: Parkinson Disease; Pain
Keywords: Parkinson Disease; Pain; tDCS; Off state; Motor fluctuations
MeSH Terms: conditions — Parkinson Disease; Pain

STUDY DESIGN:
Intervention Model Description: This study will be a triple-blinded experimental randomized controlled trial with a crossover design. The randomization will be conducted through the "GraphPad" software by an independent investigator. All the participants who fulfill the inclusion criteria and have none of the exclusion ones will be randomly allocated into two groups (depending on the order of the intervention allocation): 1.active-tDCS-2.shamtDCS or 1.sham-tDCS-2.active-tDCS. Allocation concealment will be ensured by the inclusion of the assigned group in closed opaque envelopes that will be opened at the time of the first intervention.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple-blind criteria will be achieved by identic collocation of the electrodes in both conditions and by activating the "double-blind" option in the Starstim tDCS® Software (Neuroelectrics Inc, Barcelona, Spain) that allows concealing the protocol by writing a neutral number. The evaluator, not allowed to stay in the same room while the interventions, will conceal the protocols with the neutral number and the therapist will read it in the envelope, ignoring which number coincides with each intervention. At the end of the second session, patients will be asked whether they received the order 1.active-2.sham or 1.sham-2.active, to assess the blinding success. The statistician will also be blinded through the mentioned neutral numbers. Unblinding will be permissible when any event could suppose a risk to the patient's health.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Transcranial Direct Current Stimulation and dopaminergic medication (Experimental): Active Transcranial Direct Current Stimulation (atDCS) will be applied over the Primary Motor Cortex (M1) contralateral to pain if it is unilateral, or always on the left M1 if pain is bilateral. It will consist of 1 session of 20 minutes of conventional stimulation (anode over M1) at 2 mA. It will be applied in the OFF state (i.e., >12h after the last medication intake). Lately, patients will take its usual dopaminergic medication.
  Interventions: Device: Active Transcranial Direct Current Stimulation; Device: Sham Transcranial Direct Current Stimulation; Drug: Dopaminergic medication
- : Sham Transcranial Direct Current Stimulation and dopaminergic medication (Sham Comparator): Sham Transcranial Direct Current (s-tDCS) will be applied over the Primary Motor Cortex with the same procedure, during 1 session of 20 minutes of conventional stimulation. It will be applied in the OFF state (i.e., >12h after the last medication intake). Lately, patients will take its usual dopaminergic medication.
  Interventions: Device: Active Transcranial Direct Current Stimulation; Device: Sham Transcranial Direct Current Stimulation; Drug: Dopaminergic medication

INTERVENTIONS:
Device: Active Transcranial Direct Current Stimulation — The Starstim tCS® equipment will be used, with 35 cm2 sponge electrodes. The tDCS over M1 will be performed by placing the active anode on the C3 point (10/20 EEG system) and the cathode on the contralateral supraorbital area (Fp2). Regarding the stimulated hemisphere, in cases of asymmetric pain, it will be applied to the contralateral M1, and in cases of bilateral pain, it will be applied to the M1 of the dominant hemisphere. A constant current of 2 mA (subthreshold intensity) will be applied for 20 minutes, with the first 30 seconds used as a ramp-up and the last 30 seconds as a ramp-down. Number of sessions: 1.
Device: Sham Transcranial Direct Current Stimulation — The Starstim tCS® equipment (Neuroelectrics Inc, Barcelona, Spain) will be used with 35 cm2 sponge electrodes. The tDCS sham over M1 will be performed by placing the electrodes in the same position as in the active tDCS protocol. However, the stimulator will automatically turn off after 30 seconds of stimulation, making it a reliable sham stimulation method. Therefore, subjects will feel the same tingling sensation but will not receive current for the remainder of the stimulation time.
Drug: Dopaminergic medication — After tDCS, the participant will take their regular dopaminergic medication in order to go from OFF state to ON state.

SUMMARY:
Parkinson's Disease (PD) is a neurodegenerative disorder characterized by motor and non-motor symptoms. Pain is a significant symptom in PD, affecting a large percentage of patients and impacting their quality of life. The mechanisms of pain in PD involve complex changes in pain-modulating pathways, including dopaminergic and non-dopaminergic systems.

To address the lack of pain management strategies, the investigators propose exploring non-pharmacological therapies like transcranial direct current stimulation (tDCS). tDCS is a safe and non-invasive technique that modulates neuronal activity. It has shown positive effects on pain processing in healthy individuals and chronic pain patients, but its potential for PD-associated pain remains largely unexplored.

The primary motor cortex (M1) is a target for tDCS as it is believed to influence pain processing in other brain regions involved in sensory and emotional aspects. Initial studies suggest the benefits of tDCS in PD, including enhanced motor potentials and potential modulation of dopaminergic pathways. However, there are currently no published studies specifically investigating the effects of tDCS on PD-related pain, highlighting the need for further research.

A proof-of-concept trial is proposed to examine the effects of a single tDCS session on M1 in PD patients during the OFF state (without medication) and after taking dopaminergic medication. The study aims to assess the pain-relieving effects of tDCS in PD and explore potential synergies between tDCS and dopaminergic medication. By better understanding the impact of tDCS on pain relief in PD, this research may offer insights into alternative non-pharmacological approaches for managing pain in PD.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a complex progressive neurodegenerative disorder. It is the second most common neurodegenerative disease, with a prevalence of 4.1 to 4.6 million people over the age of 50. It is estimated that these numbers will increase to 8.7 to 9.3 million by the year 2030.

PD is multisystemic and include both motor and non-motor symptoms. These symptoms can fluctuate throughout the day, leading PD patients to frequently experience two distinct states: the "on" state, when dopaminergic medication is active in their system, and the "off" state, which occurs when there is no medication concentration in the body, resulting in more severe symptoms.

Pain in PD is a highly relevant symptom that significantly impacts patients' quality of life, with a prevalence of up to 85% and moderate to severe intensity reported in 42% of individuals. Additionally, in Spain, the prevalence of PD-associated pain has significantly increased following the COVID-19 pandemic, with up to 50% of PD patients reporting daily pain. Moreover, pain in PD is often underreported, emphasizing the need to investigate its mechanisms and treatment.

The pathophysiological mechanisms of pain in PD are complex. In general, PD can lead to alterations in peripheral transmission, sensory-discriminative processing, pain perception, and interpretation at multiple levels, due to neurodegenerative changes in both dopaminergic and non-dopaminergic pain-modulating pathways. This dysregulation of the dopaminergic system can impact the experience of pain directly by enhancing nociceptive signals and indirectly by influencing expectations and the interpretation of such signals. However, it is considered that there is no specific pain center in PD patients but rather a pain matrix involving various brain structures.

Given the multiple central structures affected and their consequent pathophysiological mechanisms in PD-associated pain, there is a wide variety of clinical manifestations. These include musculoskeletal pain, generalized central chronic pain, visceral pain, pain related to "on-off" fluctuations, dystonic-dyskinetic pain, nocturnal immobility-related pain or restless legs syndrome, orofacial pain, inflammation or edema-related pain, and radicular pain.

Regarding the assessment of pain in PD, there is only one specific scale that evaluates all pain phenotypes of the disease in terms of intensity and frequency, namely the King's Parkinson's Disease Pain Scale (KPPS). Therefore, due to the scarcity of objective pain assessment tools and the crucial role of the central nervous system and endogenous modulation systems in the origin of PD-associated pain, it is important to assess pain processing characteristics such as Conditioned Pain Modulation (CPM), and Pressure Pain Thresholds (PPTs). CPM assesses the descending inhibitory pain system, and PPTs assess the intensity of pressure required to elicit initial pain in a specific body area.

Dopaminergic medication is the primary treatment for PD symptoms; however, its effects on pain management have shown contradictory results according to recent systematic reviews. Moreover, there is currently a lack of robust evidence to establish guidelines for pain management in PD, which is why non-pharmacological therapies have been proposed as a safe and useful alternative with fewer side effects.

Transcranial Direct Current Stimulation (tDCS) is a non-invasive form of brain stimulation in which a relatively weak continuous current is delivered to the cortical areas through small electrodes placed on the scalp. It is a neuromodulatory intervention, and based on the assumption that the exposed tissue is polarized, tDCS would modulate neuronal excitability by depolarizing or hyperpolarizing the resting membrane potential of neurons. This modulation would result in increases or decreases in cortical excitability, depending on whether the active electrode is the anode or the cathode, respectively.

tDCS has been shown to have an effect on certain psychophysical variables of pain processing in healthy subjects. It has primarily been shown to enhance CPM and improvements have been reported in PPTs, cold and heat pain thresholds, acute pain induced by laser (26), and pain threshold after peripheral electrical stimulation. Importantly, tDCS has also demonstrated beneficial effects in patients with chronic pain. Specifically, it has shown improvements in pain processing characteristics, resulting in clinical pain improvements in other populations with chronic neuropathic pain. It is hypothesized that tDCS could be an effective alternative in the treatment of pain with central sensitization components, a process common in PD-associated pain.

The majority of the hypoalgesic effects generated by tDCS are due to its modulation of the primary motor cortex (M1). It is suggested that tDCS over M1 could reduce pain by increasing excitability not only in the stimulated area but also in other structures involved in pain processing, both sensory and emotional, through cortico-subcortical connectivity.

However, there are currently no published studies applying tDCS for the treatment of PD-associated pain, except for unpublished studies from our group confirming a favorable effect in this regard. Nonetheless, disregarding our results, its use can be considered safe as it has already been tested in PD patients for other purposes. tDCS has demonstrated an influence on Motor Evoked Potentials (MEPs) in PD patients, increasing MEPs after stimulating M1 with an active anode and decreasing MEPs with an active cathode. Furthermore, it has been observed that bilateral tDCS with an active anode leads to increases in BDNF, thus slowing down the degeneration of dopaminergic neurons. This last piece of evidence, along with other findings that demonstrate the capacity of tDCS to modulate dopaminergic transmission, is relevant for the present project, considering that part of the descending inhibitory pain system involves these pathways. Similarly, it has been demonstrated that pain causes reductions in corticomotor excitability, governed by M1, and tDCS applied to M1 has shown the ability to increase cortical excitability, which has abnormal activity in PD patients and could influence their pain.

Given the overlap between many influential areas in PD-associated pain and the areas excited by tDCS over M1, with these increases in excitability correlating with pain reduction, as well as the potential effect of tDCS on dopaminergic pathways, a hypoalgesic effect of tDCS in PD patients in their OFF state is hypothesized. Additionally, if the action is based on the activation of dopaminergic pathways, a possible enhancement of dopaminergic medication's action with better pain control during the ON period is also expected. However, there is currently no study that has specifically evaluated this effect in PD patients in the OFF state, making it pertinent to conduct a proof-of-concept trial with this objective. The objective is to determine the effect of a single session of treatment using transcranial direct current stimulation (tDCS) on the primary motor cortex (M1) on perceived clinical pain and pain processing characteristics in patients with Parkinson's disease (PD) in the OFF state (without dopaminergic medication) and after taking dopaminergic medication.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Idiopathic Parkinson´s Disease.
* Presence of Parkinson´s Disease-related pain in the off-state.
* Neuroimaging study without previous pathologies.
* Score > 5 in transfers (bed to chair and back) item in Barthel Index.
* Score = or > 26 in Montreal Cognitive Assessment (MoCA).
* Tolerability for the application of electrotherapy.
* Able to provide informed consent to participate in the study
* Pain intensity >= 3 in Visual Analogue Scale or equivalent.

Exclusion Criteria:

* Neurologic disease different from PD.
* Pain non-related to PD.
* Dermatologic problems, wounds, or ulcers in the electrode's application area.
* Presence of implants or metal pieces in the head.
* Presence of cardiac pacemaker, vagal, brain or transcutaneous stimulators, medication pumps, ventriculoperitoneal shunts or aneurysm clips.
* Significative difficulties in language.
* History of alcohol or drugs abuse.
* Non-controlled medical problems.
* Pregnancy.
* Epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Change in Conditioned Pain Modulation | From baseline to immediately post tDCS
  Assesses the descending pain modulatory system. The Pain Pressure Threshold will be assessed in the middle ofthe distal phalanx of the thumb with ta handheld algometer, corresponding to the first test stimulus. Afterward, the patient will immerse the contrary hand up to the wrist into stirred ice-cold water (0-4º) maintaining it for 3 minutes, corresponding to the conditioning stimulus. If the pain is unbearable before the 3 minutes, the patient will be able to remove his/her hand. Immediately after removing the hand, a second Pain Pressure Threshold measure will be performed in the same place as the first one, corresponding to the second test stimulus. After 1-minute rest, a third Pain Pressure Threshold will be measured to assess the Conditioned Pain Modulation residual functioning.
Change in Conditioned Pain Modulation | From baseline to immediately post dopaminergic medication
  Assesses the descending pain modulatory system. The Pain Pressure Threshold will be assessed in the middle ofthe distal phalanx of the thumb with ta handheld algometer, corresponding to the first test stimulus. Afterward, the patient will immerse the contrary hand up to the wrist into stirred ice-cold water (0-4º) maintaining it for 3 minutes, corresponding to the conditioning stimulus. If the pain is unbearable before the 3 minutes, the patient will be able to remove his/her hand. Immediately after removing the hand, a second Pain Pressure Threshold measure will be performed in the same place as the first one, corresponding to the second test stimulus. After 1-minute rest, a third Pain Pressure Threshold will be measured to assess the Conditioned Pain Modulation residual functioning.
Changes in Pain Pressure Threshold | From baseline to immediately post tDCS
  Two Pain Pressure Thresholds will be measured by a handheld algometer, one over the most painful area (peripheric hyperalgesia) and the other one over the middle of the distal phalanx of the thumb (central hyperalgesia). The Pain Pressure Threshold will be applied with the algometer perpendicular to the skin increasing at a rate of 1 kg/s until the first sensation of pain. 3 measures with 30-seconds rest between pulses will be performed, taking the average as Pain.
  Pressure Threshold.
Changes in Pain Pressure Threshold | From baseline to immediately post dopaminergic medication
  Two Pain Pressure Thresholds will be measured by a handheld algometer, one over the most painful area (peripheric hyperalgesia) and the other one over the middle of the distal phalanx of the thumb (central hyperalgesia). The Pain Pressure Threshold will be applied with the algometer perpendicular to the skin increasing at a rate of 1 kg/s until the first sensation of pain. 3 measures with 30-seconds rest between pulses will be performed, taking the average as Pain.
  Pressure Threshold.
Changes in Visual Numeric Pain Rating Scale | From baseline to immediately post tDCS
  It will be used to measure pain intensity due to its high discriminatory power. The scale assesses pain intensity using numbers or words through various types of scales ranging from 0 to 10. Pain rating ranges from 0 (no pain), 1-3 (mild pain, mild discomfort or irritation, slight impairment in daily activities), 4-6 (moderate pain, significant impairment in daily activities), and 7-10 (severe pain, inability to perform daily activities).
Changes in Visual Numeric Pain Rating Scale | From baseline to immediately post dopaminergic medication
  It will be used to measure pain intensity due to its high discriminatory power. The scale assesses pain intensity using numbers or words through various types of scales ranging from 0 to 10. Pain rating ranges from 0 (no pain), 1-3 (mild pain, mild discomfort or irritation, slight impairment in daily activities), 4-6 (moderate pain, significant impairment in daily activities), and 7-10 (severe pain, inability to perform daily activities).
Changes in Global Rating of Change | From baseline to immediately post tDCS
  It will be used to measure the self-perceived change in the patient's pain state. Its main objective is to quantify the extent to which a patient has improved or worsened over a specific period of time. It involves a single question asked to the patient to rate their change compared to the pre-intervention state, and the scores will range from -7 (much worse than before), through 0 (same as before), to +7 (much better than before).
Changes in Global Rating of Change | From baseline to immediately post dopaminergic medication
  It will be used to measure the self-perceived change in the patient's pain state. Its main objective is to quantify the extent to which a patient has improved or worsened over a specific period of time. It involves a single question asked to the patient to rate their change compared to the pre-intervention state, and the scores will range from -7 (much worse than before), through 0 (same as before), to +7 (much better than before).

SECONDARY OUTCOMES:
Changes in Brain Symmetry Index in electroencephalography | From baseline to immediately post tDCS
  Resting state EEG: A 64-channel EEG recording will be performed at rest for 3 minutes following the standard protocol for baseline assessment.
  Tapping EEG: A 64-channel EEG recording will be conducted while performing a tapping task for 30 seconds. The recording will be done separately for each hand, starting with the dominant hand.
  Closed-Eyes EEG: A 64-channel EEG recording will be conducted while participants have their eyes closed for 5 minutes.
Changes in Brain Symmetry Index in electroencephalography | From baseline to immediately post dopaminergic medication
  Resting EEG: A 64-channel EEG recording will be performed at rest for 3 minutes following the standard protocol for baseline assessment.
  Tapping EEG: A 64-channel EEG recording will be conducted while performing a tapping task for 30 seconds. The recording will be done separately for each hand, starting with the dominant hand.
  Closed-Eyes EEG: A 64-channel EEG recording will be conducted while participants have their eyes closed for 5 minutes.
Changes in Unified Parkinson´s Disease Rating Scale | From baseline to immediately post dopaminergic medication
  It is a quantitative scale that collects information about the frequency and severity of motor symptoms. Higher scores indicate a greater degree of impairment. The minumum value is 0 and the maximum is 68.
Changes in Finger tapping task | From baseline to immediately post dopaminergic medication
  Finger Taping task, where the participants will be instructed to press the space bar on the keyboard as fast as possible and repeatedly with the index finger, to measure motor function.

OTHER OUTCOMES:
King´s Parkinson´s Disease Pain Scale score | Baseline
  Parkinson´s Disease specific scale that evaluates the localization, frequency, and intensity of pain. It has 14 items distributed in 7 domains: 1. Musculoskeletal Pain; 2. Chronic Pain; 3. Fluctuation-related Pain; 4. Nocturnal Pain; 5. Oro-facial Pain; 6. Discoloration, Oedema/Swelling Pain; 7. Radicular Pain. Each item is scored by severity (0, none to 3, very severe) multiplied by frequency (0, never to 4, all the time) resulting in a subscore of 0 to 12, the sum of which gives the total score with a theoretical range from 0 to 168, with higher scores indicating more severity and frequency of pain.
Brief Pain Inventory score | Baseline
  It contains 15 items, including 2 multi-item scales to measure the intensity of pain and its impact on the function and welfare of patients. It also presents open questions to assess the localization of pain and the treatment used for its management, just as its effectiveness. Scores oscillate from 0 to 110, with higher scores indicating more pain and more impact on function and welfare of patients
Beck´s Depression Inventory | Baseline
  Measures depressive symptoms. Scores range from 0 to 63 leading to 6 groups: 0-10, normal; 11-16, mild mood disturbance; 17-20, borderline clinical depression; 21-30, moderate depression; 31-40, severe depression; and over 40, extreme depression
State-Trait Anxiety Inventory | Baseline
  Measures anxious states and anxious traits. It has 20 items for assessing trait anxiety and 20 for state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety
Tampa Scale of Kinesiophobia | Baseline
  Measures fear of movement-related pain. Its scores range from 11-44 points with higher scores indicating greater fear of pain, movement, and injury
Pain Catastrophizing Scale | Baseline
  Measures catastrophizing thinking. Its total score range from 0-52, along with three subscale scores assessing rumination, magnification and helplessness, with higher scores indicating higher level of catastrophizing.
PD-specific 16-items Parkinson Fatigue Scale | Baseline
  It is a scale that measures the specific fatigue experienced by patients with Parkinson's disease. It consists of 16 items with five response categories ranging from 0 (strongly disagree) to 4 (strongly agree). The final sum of these items yields a total score ranging from zero to 64, with higher scores indicating higher levels of fatigue. If the scale is not available in Spanish, either the Fatigue Severity Scale (FSS) or the Multidimensional Fatigue Inventory (MFI) will be used, as they have been validated for Parkinson's disease and recommended by the International Parkinson and Movement Disorder Society (MDS).

CONTACTS AND LOCATIONS:
Overall Officials: Juan Pablo Romero, MD, PhD, Principal Investigator — Universidad Francisco de Vitoria, Facultad de Ciencias Experimentales; Josué Fernández Carnero, PT, PhD, Principal Investigator — Universidad Rey Juan Carlos; Marcos Moreno Verdú, PT, PhD, Principal Investigator — Universidad Francisco de Vitoria
Locations (1):
- Hospital Beata Maria Ana, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual anonymized participant data will be available to other researchers under request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Four months at the end of the study
Access Criteria: Individual anonymized participant data will be available to other researchers under request.

REFERENCES:
- [Result] Kalia LV, Lang AE. Parkinson's disease. Lancet. 2015 Aug 29;386(9996):896-912. doi: 10.1016/S0140-6736(14)61393-3. Epub 2015 Apr 19. PMID 25904081
- [Result] Silverdale MA, Kobylecki C, Kass-Iliyya L, Martinez-Martin P, Lawton M, Cotterill S, Chaudhuri KR, Morris H, Baig F, Williams N, Hubbard L, Hu MT, Grosset DG; UK Parkinson's Pain Study Collaboration. A detailed clinical study of pain in 1957 participants with early/moderate Parkinson's disease. Parkinsonism Relat Disord. 2018 Nov;56:27-32. doi: 10.1016/j.parkreldis.2018.06.001. Epub 2018 Jun 6. PMID 29903584
- [Result] Antonini A, Tinazzi M, Abbruzzese G, Berardelli A, Chaudhuri KR, Defazio G, Ferreira J, Martinez-Martin P, Trenkwalder C, Rascol O. Pain in Parkinson's disease: facts and uncertainties. Eur J Neurol. 2018 Jul;25(7):917-e69. doi: 10.1111/ene.13624. Epub 2018 Apr 18. PMID 29520899
- [Result] Lefaucheur JP, Antal A, Ayache SS, Benninger DH, Brunelin J, Cogiamanian F, Cotelli M, De Ridder D, Ferrucci R, Langguth B, Marangolo P, Mylius V, Nitsche MA, Padberg F, Palm U, Poulet E, Priori A, Rossi S, Schecklmann M, Vanneste S, Ziemann U, Garcia-Larrea L, Paulus W. Evidence-based guidelines on the therapeutic use of transcranial direct current stimulation (tDCS). Clin Neurophysiol. 2017 Jan;128(1):56-92. doi: 10.1016/j.clinph.2016.10.087. Epub 2016 Oct 29. PMID 27866120
- [Result] Fregni F, Boggio PS, Santos MC, Lima M, Vieira AL, Rigonatti SP, Silva MT, Barbosa ER, Nitsche MA, Pascual-Leone A. Noninvasive cortical stimulation with transcranial direct current stimulation in Parkinson's disease. Mov Disord. 2006 Oct;21(10):1693-702. doi: 10.1002/mds.21012. PMID 16817194
- [Result] Fregni F, Boggio PS, Lima MC, Ferreira MJ, Wagner T, Rigonatti SP, Castro AW, Souza DR, Riberto M, Freedman SD, Nitsche MA, Pascual-Leone A. A sham-controlled, phase II trial of transcranial direct current stimulation for the treatment of central pain in traumatic spinal cord injury. Pain. 2006 May;122(1-2):197-209. doi: 10.1016/j.pain.2006.02.023. Epub 2006 Mar 27. PMID 16564618
- [Result] Chaudhuri KR, Rizos A, Trenkwalder C, Rascol O, Pal S, Martino D, Carroll C, Paviour D, Falup-Pecurariu C, Kessel B, Silverdale M, Todorova A, Sauerbier A, Odin P, Antonini A, Martinez-Martin P; EUROPAR and the IPMDS Non Motor PD Study Group. King's Parkinson's disease pain scale, the first scale for pain in PD: An international validation. Mov Disord. 2015 Oct;30(12):1623-31. doi: 10.1002/mds.26270. Epub 2015 Jun 11. PMID 26096067
- [Result] Perez-Lloret S, Ciampi de Andrade D, Lyons KE, Rodriguez-Blazquez C, Chaudhuri KR, Deuschl G, Cruccu G, Sampaio C, Goetz CG, Schrag A, Martinez-Martin P, Stebbins G; Members of the MDS Committee on Rating Scales Development. Rating Scales for Pain in Parkinson's Disease: Critique and Recommendations. Mov Disord Clin Pract. 2016 Jun 24;3(6):527-537. doi: 10.1002/mdc3.12384. eCollection 2016 Nov-Dec. PMID 30363588
- [Result] Imai Y, Petersen KK, Morch CD, Arendt Nielsen L. Comparing test-retest reliability and magnitude of conditioned pain modulation using different combinations of test and conditioning stimuli. Somatosens Mot Res. 2016 Sep-Dec;33(3-4):169-177. doi: 10.1080/08990220.2016.1229178. Epub 2016 Sep 20. PMID 27650216
- [Result] Santos-Garcia D, Oreiro M, Perez P, Fanjul G, Paz Gonzalez JM, Feal Painceiras MJ, Cores Bartolome C, Valdes Aymerich L, Garcia Sancho C, Castellanos Rodrigo MDM. Impact of Coronavirus Disease 2019 Pandemic on Parkinson's Disease: A Cross-Sectional Survey of 568 Spanish Patients. Mov Disord. 2020 Oct;35(10):1712-1716. doi: 10.1002/mds.28261. Epub 2020 Sep 22. PMID 32776601
- [Derived] Gonzalez-Zamorano Y, Moreno-Verdu M, Martinez-Benito A, Fernandez-Carnero J, Romero JP. Transcranial Direct Current Stimulation in Parkinson's Disease Patients in the Off State: A Randomized Controlled Crossover Trial Examining the Effects on Pain With and Without the Influence of Dopaminergic Medication. Pain Pract. 2025 Nov;25(8):e70082. doi: 10.1111/papr.70082. PMID 41039704